CLINICAL TRIAL: NCT02170506
Title: Effect of Sub-mental Sensitive Transcutaneous Electrical Stimulation on Pharyngeal Muscles Control
Brief Title: Effect of Sub-mental Sensitive Transcutaneous Electrical Stimulation on Pharyngeal Muscles Control : TENSVIRT Study
Acronym: TENSVIRT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Rouen (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: 2013/176/HP
Record Dates: First submitted 2014-03-19; First posted 2014-06-23 (Estimated); Last update posted 2015-01-22 (Estimated); Status verified 2015-01

CONDITIONS: Oropharyngeal Dysphagia; Deglutition Disorders
MeSH Terms: conditions — Deglutition Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- submental sensitive transcutaneous electrical stimulation. (Experimental): Each Healthy subjects will be his own witness. Urostim 2 stimulation Arm
  Interventions: Device: Urostim 2 stimulation

INTERVENTIONS:
Device: Urostim 2 stimulation — Sensory transcutaneous electrical stimulation will be started for a period of 20 minutes. It is applied by means of two surface electrodes placed under chin stimulation of both sides of the center line of the preceding side. Sensory transcutaneous electrical stimulation will inhibit the cerebral control of swallowing.
  Other Names: Device transcutaneous neuromuscular electrical stimulation

SUMMARY:
Swallowing is a complex phenomenon that allows oral feeding while protecting the airway. It involves many brain areas, including primary motor and sensory areas. Its dysfunction, called oropharyngeal dysphagia is present in approximately 60% of patients with a stroke. In this case, it is conventionally translated by a swallow response time delay of the swallowing reflex.

Pathophysiology of dysphagia is explained by impairment of the dominant swallowing, function that representation center is bi-hemispheric but asymmetric (Hamdy, 1997). Half of patients with a stroke supra-tentoriel with oropharyngeal dysphagia (about 55 % of strokes) regain normal swallowing in a few weeks ( Barer, 1989). Mechanisms that determine the recovery appear to be related to a reorganization of the motor cortex intact. Patients who retain disorders are those who have not cortical reorganization.

With this in mind a team used different methods known to modulate brain plasticity, which electrotherapy with an application endo- pharyngeal sensory threshold. This stimulation increases the excitability of the cortico- bulbar reflex, which improves swallowing function in the clinical application.

The hypothesis of this work is that the transcutaneous electrical stimulation applied submental, noninvasive technique, would also have an impact on cortical plasticity may explain the improved coordination of swallowing observed in earlier studies (Verin , 2011) ( Gallas , 2010).

ELIGIBILITY:
Inclusion Criteria:

1. Subjects aged over 18 years
2. Affilitation to social security scheme
3. Registration in National register of people who participate in biomedical research
4. Healthy volunteers who provided written informed consent

Exclusion Criteria:

1. Subjects with swallowing disorders
2. Presence of psychiatric disorders
3. Skin disorders
4. Cardiac disorders (non controlled arrythmia, severe heart failure, presence of heart valve)
5. Submental tumor
6. Epilepsia, treated or untreated
7. Presence of neurosurgical clip
8. Suspicion of digestive fistula
9. Presence of metal, pacemaker, defibrillator, pump treatment or neurostimulation
10. Cannabis user, regular use of benzodiazepines
11. Presence of chronic respiratory, neurological disease, ENT or gastroesophageal disease (cause potentially change swallowing)
12. Contra-indication to MRI (claustrophobia, metal fragment, cardiac/ENT/neurological implantable device not MRI compatible, osteosynthesis prior to 1980)
13. Subject reported against the use of Micropaque®
14. Pregnant or nursing woman, or absence of contraception
15. Poor understanding of French langage
16. Person under judicial protection
17. Person deprive of their liberty by judicial or administrative decision
18. Participating in a clinical trial within 4 weeks before the pre-inclusion visit

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2014-04; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Variation in motor evoked potential amplitude | 1 month
  Our aim was to show that submental sensitive transcutaneous electrical stimulation (SSTES) can modified swallowing function. Primary endpoint is change in motor evoked potential amplitude after submental transcutaneous electrical stimulation

SECONDARY OUTCOMES:
variation of swallow reaction time | 1 Month
  highlighting a change in swallowing with videofluoroscopy studied with electrical stimulation. Secondary endpoints are :
  * modification of swallowing cortical area
  * variation of swallow reaction time on videofluoroscopy

CONTACTS AND LOCATIONS:
Overall Officials: Eric VERIN, Professor, Principal Investigator — University Hospital, Rouen
Locations (1):
- UHRouen, Rouen, France